CLINICAL TRIAL: NCT06430944
Title: Comparative Study Between Single and Double Limb Hip Spica Cast in Fracture Femur in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS-318-2023
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Femur Fracture
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single limb spica casting: (Experimental): A folded towel was placed inside the tubular bandage over the centre of the abdomen, which helped create breathing space inside the cast. The towel's tail was brought towards the neck for easier removal.
  Then, a layer of the padded cast was applied using a large width for the body and a narrower one for the lower limb. A thick felt was added over this padding along the free edges of the chest and the leg. The first layer of the cast was applied to the leg and body in an eight-figure manner, taking care to connect the leg to the body securely. The reinforced cast slabs were applied between the body and the lower limb segments. The thigh segment was moulded to maintain a good reduction by keeping the anterolateral of the cast flat or slightly concave. Some clinicians moulded the segment enough to result in ten degrees of initial valgus.
  Interventions: Procedure: Placing a hip spica cast for patients with femur fractures
- Double limb spica cast: (Active Comparator): One and a half cast was applied in a single limb spica cast, extending to the opposite leg to the knee. Reinforced slabs were applied to hip joints in both limbs
  Interventions: Procedure: Placing a hip spica cast for patients with femur fractures

INTERVENTIONS:
Procedure: Placing a hip spica cast for patients with femur fractures — Placing a hip spica cast for patients with femur fractures. These hip spicas are made for each patient to stabilize the fracture in pediatric patients

SUMMARY:
We performed a randomized control trial including 84 children aged two to six years who presented with femoral fractures. They were randomized into two groups; the first was managed by single limb cast fixation (42 patients), and the second was managed by double limb cast fixation (42 patients). The primary outcomes were postprocedural functional outcomes and parents' satisfaction, while the secondary outcomes were the rates of complications.

DETAILED DESCRIPTION:
Femoral fractures are frequent in children and compose 1% to 2% of all pediatric fractures. Conservative management is associated with good results, whether by single or double-limb cast fixations. We aim to compare both procedures regarding functional outcomes, complications, and parents' satisfaction. Eighty-four children were eligible to be included in our study; 42 underwent single limb spica casts, and the other 42 patients underwent double limb spica casts. Both groups had similar baseline characteristics like age, gender, fracture side, and fracture classification.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 to 6 years
* Children with femur shaft fractures

Exclusion Criteria:

* Children younger than 2 years or older than 6 years
* Articular fractures or fractures that cant be managed with a cast
* Old fractures older than 3 weeks

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Flynn's score | 6 months
  The Flynn evaluation system is based on the presence of leg length inequality, malalignment, pain, and minor and major complications. Each of these criteria is either defined as Excellent, successful or poor.

SECONDARY OUTCOMES:
loss of reduction | 6 months
  we do xrays to confirm if there is any loss of reduction of the fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy-Cairo University- Faculty of Medicine, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided